CLINICAL TRIAL: NCT06722729
Title: A Late Phase II Clinical Trial of KDT-3594 in Patients With Advanced Parkinson's Disease With Levodopa
Brief Title: A Late Phase II Clinical Trial of KDT-3594 in Patients With Parkinson's Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KDT1203; Under registration (Registry Identifier: jRCT)
Record Dates: First submitted 2024-11-26; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-11

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KDT-3594 (Experimental): KDT-3594 capsules will be orally administered at escalating doses ranging from 0.25 to 2 mg per day for 17 weeks.
  Interventions: Drug: KDT-3594
- Placebo (Placebo Comparator): Placebo capsules will be orally administered at escalating doses ranging from 0.25 to 2 mg per day for 17 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KDT-3594 — Oral administration
  Arms: KDT-3594
Drug: Placebo — Oral administration
  Arms: Placebo

SUMMARY:
This trial is a late phase II, multicenter, randomized, double-blind, placebo-controlled, parallel group trial to evaluate the efficacy, safety, and pharmacokinetics of KDT-3594 administered at escalating doses ranging from 0.25 to 2 mg per day for 17 weeks in patients with advanced PD with levodopa.

DETAILED DESCRIPTION:
This trial is a late phase II, multicenter, randomized, double-blind, placebo-controlled, parallel group trial to evaluate the efficacy, safety, and pharmacokinetics of KDT-3594 administered once daily in patients with advanced PD with levodopa.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with PD according to the Parkinson's disease society brain bank clinical diagnostic criteria of the UK Parkinson's Disease Society
* Patients who are being treated with levodopa or levodopa combination drugs and have any of the following troublesome symptoms or conditions:
* Patients with wearing-off phenomenon
* Patients with ON-/OFF-phenomenon
* Patients with no-on/delayed on phenomenon
* Patients with inadequate response to levodopa

Exclusion Criteria:

* Patients suspected of having parkinsonism other than PD based on medical history, physical findings, laboratory test values, dopamine transporter-single photon emission computed tomography (DAT-SPECT), etc.
* Patients who have undergone neurosurgical therapy for PD (e.g., stereotactic thalamotomy and pallidotomy and deep brain stimulation) or who are scheduled to undergo surgical therapy during the trial period
* Patients complicated with overt dementia or a Mini-Mental State Examination (MMSE) score of < 24 at the start of the screening period

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the MDS-UPDRS Part II+III (ON-time) total score at Week 17 of the treatment period | Up to 17 weeks
  MDS-UPDRS is a multimodal scale assessing impairment and disability consisting of 4 parts. (Part I; 13 items) non-motor experiences of daily living, (Part II; 13 items) motor experiences of daily living completed by the participants, (Part III; 33 items) motor examination of PD and was administered by the rater, and (Part IV; 6 items) motor complication integrates participant-derived information with the rater's clinical observations and judgements and is completed by the rater. For each question, a numeric score was assigned between 0-4, where 0 = Normal, 1 = Slight, 2 = Mild, 3 = Moderate, 4 = Severe. In all parts, a higher score indicated more severe symptoms of PD, and the score range of each part are as follows.
  * Part I: 0-52
  * Part II: 0-52
  * Part III: 0-132
  * Part IV: 0-24
  * Total Score: 0-260
  * Part II+III: 0-184 (MDS-UPDRS Part II and III combined score equals the sum of Parts II and III (range 0-184)).

SECONDARY OUTCOMES:
Change from baseline in the MDS-UPDRS Part II+III (ON-time) total score | Up to 17 weeks
  MDS-UPDRS is a multimodal scale assessing impairment and disability consisting of 4 parts. (Part I; 13 items) non-motor experiences of daily living, (Part II; 13 items) motor experiences of daily living completed by the participants, (Part III; 33 items) motor examination of PD and was administered by the rater, and (Part IV; 6 items) motor complication integrates participant-derived information with the rater's clinical observations and judgements and is completed by the rater. For each question, a numeric score was assigned between 0-4, where 0 = Normal, 1 = Slight, 2 = Mild, 3 = Moderate, 4 = Severe. In all parts, a higher score indicated more severe symptoms of PD, and the score range of each part are as follows.
  * Part I: 0-52
  * Part II: 0-52
  * Part III: 0-132
  * Part IV: 0-24
  * Total Score: 0-260
  * Part II+III: 0-184 (MDS-UPDRS Part II and III combined score equals the sum of Parts II and III (range 0-184)).
Change from baseline in the MDS-UPDRS Part I, II, III, and IV (ON-time) total score | Up to 17 weeks
  MDS-UPDRS is a multimodal scale assessing impairment and disability consisting of 4 parts. (Part I; 13 items) non-motor experiences of daily living, (Part II; 13 items) motor experiences of daily living completed by the participants, (Part III; 33 items) motor examination of PD and was administered by the rater, and (Part IV; 6 items) motor complication integrates participant-derived information with the rater's clinical observations and judgements and is completed by the rater. For each question, a numeric score was assigned between 0-4, where 0 = Normal, 1 = Slight, 2 = Mild, 3 = Moderate, 4 = Severe. In all parts, a higher score indicated more severe symptoms of PD, and the score range of each part are as follows.
  * Part I: 0-52
  * Part II: 0-52
  * Part III: 0-132
  * Part IV: 0-24
  * Total Score: 0-260
  * Part II+III: 0-184 (MDS-UPDRS Part II and III combined score equals the sum of Parts II and III (range 0-184)).
Response rate in the MDS-UPDRS Part III (ON-time) total score | Up to 17 weeks
  MDS-UPDRS is a multimodal scale assessing impairment and disability consisting of 4 parts. (Part I; 13 items) non-motor experiences of daily living, (Part II; 13 items) motor experiences of daily living completed by the participants, (Part III; 33 items) motor examination of PD and was administered by the rater, and (Part IV; 6 items) motor complication integrates participant-derived information with the rater's clinical observations and judgements and is completed by the rater. For each question, a numeric score was assigned between 0-4, where 0 = Normal, 1 = Slight, 2 = Mild, 3 = Moderate, 4 = Severe. In all parts, a higher score indicated more severe symptoms of PD, and the score range of each part are as follows.
  * Part I: 0-52
  * Part II: 0-52
  * Part III: 0-132
  * Part IV: 0-24
  * Total Score: 0-260
  * Part II+III: 0-184 (MDS-UPDRS Part II and III combined score equals the sum of Parts II and III (range 0-184)).
Change from baseline in the proportion of OFF-time in awake time | Up to 17 weeks
Change from baseline in OFF-time | Up to 17 weeks
Incidence of adverse events and treatment-related adverse events | Up to 17 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yoshitaka Shimizu, Study Director — Kissei Pharmaceutical Co., Ltd.
Locations (1):
- Research Site, Multiple Locations, Japan

IPD SHARING:
Plan to Share IPD: No